CLINICAL TRIAL: NCT04760899
Title: Bilateral Cerebellar Transcranial Direct Current Stimulation (tDCS) for the Treatment of Sports-Related Post-Concussion Syndrome (SRPCS)
Brief Title: Cerebellar TDCS for SRPCS Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Justin Deters, Principal Investigator, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202011163
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Post-Concussion Syndrome
MeSH Terms: conditions — Post-Concussion Syndrome | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Active Group (Active Comparator): This group will receive the active form of tDCS. The tDCS will be administered with the anode over the right lobule of the cerebellum, and the cathode over the left lobule of the cerebellum. Stimulation will be administered for a twenty minute period that does not include the 30 second ramp up at the beginning and end of the stimulation.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham Group (Sham Comparator): This group will receive the sham form of tDCS. The electrodes will be placed in the same montage as in the Active group, however the stimulation parameters are different. For this group, the stimulation will be ramped up to the target intensity over thirty seconds at the beginning, then immediately ramp down over thirty seconds. The stimulation will then remain off for the next twenty minutes. After twenty minutes the stimulation will ramp up to the target intensity and then back down over thirty seconds.
  Interventions: Device: Transcranial Direct Current Stimulation
- Healthy Controls (No Intervention): These will be age and sex-matched healthy controls who only come in for the baseline visit in order to provide comparative values with which to confirm adequate impairment in our diseased population.

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation is a form of non-invasive brain stimulation. It uses small electrodes to deliver small amounts of current to specific areas of the brain to either increase or decrease excitability.
  Other Names: tDCS
  Arms: Active Group; Sham Group

SUMMARY:
This study is investigating the immediate and long-term effects of bilateral cerebellar transcranial direct current stimulation on cognition, balance, and symptom severity in people with sports-related post-concussion syndrome. The central hypothesis is that tDCS will provide improvements in cognitive deficits, balance, and overall symptom attenuation in people with SRPCS both acutely and at 2 and 4 week follow ups. The researchers further hypothesize that cerebellar tDCS will ameliorate the symptoms of people with SRPCS.

DETAILED DESCRIPTION:
The long term goal is to develop an effective and broadly applicable treatment modality for athletes who develop SPRCS. The objective of this study is to investigate the effects of multiple (5 consecutive daily) sessions of 2 milliampere (mA) right cerebellar tDCS on cognitive deficits, balance, and overall attenuation of symptoms on people with SRPCS. Cognitive deficits will be assessed with the N-back Working Memory test, list sorting test, and dimensional change card test. Balance deficits will be assessed with the Berg Balance Scale and Standing Balance Test (SBT), and symptoms will be assessed via the Rivermead Post-Concussion Symptom Questionnaire (RPQ). The cognitive and balance tasks are taken from the NIH motor toolbox and have been shown to be the most important for health and success in school and work, and the RPQ is one of the most widely used SRPCS evaluation tools. The central hypothesis is that tDCS will provide improvements in cognitive deficits, balance, and overall symptom attenuation in people with SRPCS both acutely and at 2 and 4 week follow ups. The researchers further hypothesize that cerebellar tDCS will ameliorate the symptoms of people with SRPCS. The rationale is that the results will improve the quality of life of these patients and may prevent impairment of cognitive function later in life.

ELIGIBILITY:
Inclusion Criteria:

1. Sign Informed Consent Document
2. Stated willingness to comply with all study procedures and availability for the duration of the study Male or female, aged 18-30.
3. Diagnosed with a concussion by a doctor greater than or equal to 1 month ago.
4. Concussion occurring during a sport/recreational activity
5. Meet the ICD-10 diagnostic criteria for Post Concussion Syndrome:

   1. history of a traumatic brain injury at least a month in the past
   2. 3 or more of the following symptoms: headaches, dizziness, fatigue, irritability, insomnia, concentration, memory difficulty
6. Rivermead Post Concussion Questionnaire score of at least 21 at baseline.
7. Comprehension of the protocol, as indicated by an ability to respond to questions about the study after reading the consent form.
8. Healthy enough to complete the protocol based, on information obtained from a clinical exam and past medical history.
9. Able to use and be contacted by telephone
10. Able to speak, read, and understand English, and complete questionnaires in English.

Healthy Controls

1. No history of mild traumatic brain injury or diagnosed concussion within the last year.
2. Not suffering from any PCS symptoms related to a brain injury
3. No History of a psychiatric condition (other than mild to moderate anxiety or depression)
4. Currently on no prescribed psychoactive medications
5. Comprehension of the protocol, as indicated by an ability to respond to questions about the study after reading the consent form.
6. Healthy enough to complete the protocol based, on information obtained from a clinical exam and past medical history.
7. Able to use and be contacted by telephone
8. Able to speak, read, and understand English, and complete questionnaires in English

Exclusion Criteria:

- 1. History/presence of secondary conditions such as seizure disorders (or on medications known to lower seizure threshold), hydrocephalus, diabetes mellitus, or claustrophobia 2. Currently diagnosed drug and/or alcohol addiction 3. Active Psychosis 4. History of a psychiatric condition (other than mild to moderate anxiety or depression) 5. Currently on no prescribed psychoactive medications 6. Not in any kind of memory improvement program or therapy during study participation.

7. Pregnancy 8. No known fissures or holes in the skull 9. No metallic objects or implanted devices in the skull

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | 2 weeks
  Balance Assessment. This is a 14 item test with scores from 0 to 4, with 4 being no inhibition at all. The max score on this test is 56, higher scores indicating better balance.
Standing Balance Test | 2 weeks
  Balance Assessment. Outcomes of this test are overall postural sway translated into a normalized t-score.
Flanker Inhibitory Control Test | 2 weeks
  Assessment of Cognition/
Dimensional Change Card Sorting Test | 2 weeks
  Assessment of Cognition
List Sorting Working Memory Test | 2 weeks
  Assessment of Cognition

SECONDARY OUTCOMES:
Dimensional Change Card Sorting Test | 2 and 4 week follow ups
  Assessment of Cognition
Berg Balance Scale | 2 and 4 week follow ups
  Balance Assessment. This is a 14 item test with scores from 0 to 4, with 4 being no inhibition at all. The max score on this test is 56, higher scores indicating better balance.
Standing Balance Scale | 2 and 4 week follow ups
  Balance Assessment. Outcomes of this test are overall postural sway translated into a normalized t-score.
Flanker Inhibitory Control Test | 2 and 4 week follow ups
  Assessment of Cognition
List Sorting Working Memory Test | 2 and 4 week follow ups
  Assessment of Cognition

CONTACTS AND LOCATIONS:
Locations (1):
- Thorsten of Rudroff, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conder A, Conder R, Friesen C. Neurorehabilitation of Persistent Sport-Related Post-Concussion Syndrome. NeuroRehabilitation. 2020;46(2):167-180. doi: 10.3233/NRE-192966. PMID 32083597
- [Background] DePadilla L, Miller GF, Jones SE, Peterson AB, Breiding MJ. Self-Reported Concussions from Playing a Sport or Being Physically Active Among High School Students - United States, 2017. MMWR Morb Mortal Wkly Rep. 2018 Jun 22;67(24):682-685. doi: 10.15585/mmwr.mm6724a3. PMID 29927909
- [Background] Doroszkiewicz C, Gold D, Green R, Tartaglia MC, Ma J, Tator CH. Anxiety, Depression, and Quality of Life: A Long-Term Follow-Up Study of Patients with Persisting Concussion Symptoms. J Neurotrauma. 2021 Feb 15;38(4):493-505. doi: 10.1089/neu.2020.7313. Epub 2020 Nov 2. PMID 32962513
- [Background] Eagle SR, Kontos AP, Collins MW, Connaboy C, Flanagan S. Network Analysis of Sport-related Concussion Research During the Past Decade (2010-2019). J Athl Train. 2020 Nov 5. doi: 10.4085/280-20. Online ahead of print. PMID 33150356
- [Background] Chen CL, Lin MY, Huda MH, Tsai PS. Effects of cognitive behavioral therapy for adults with post-concussion syndrome: A systematic review and meta-analysis of randomized controlled trials. J Psychosom Res. 2020 Sep;136:110190. doi: 10.1016/j.jpsychores.2020.110190. Epub 2020 Jul 17. PMID 32712533
- [Background] Willer B, Leddy JJ. Management of concussion and post-concussion syndrome. Curr Treat Options Neurol. 2006 Sep;8(5):415-26. doi: 10.1007/s11940-006-0031-9. PMID 16901381
- [Background] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Background] Demirtas-Tatlidede A, Vahabzadeh-Hagh AM, Bernabeu M, Tormos JM, Pascual-Leone A. Noninvasive brain stimulation in traumatic brain injury. J Head Trauma Rehabil. 2012 Jul-Aug;27(4):274-92. doi: 10.1097/HTR.0b013e318217df55. PMID 21691215
- [Background] Laidi C, Levenes C, Suarez-Perez A, Fevrier C, Durand F, Bouaziz N, Januel D. Cognitive Impact of Cerebellar Non-invasive Stimulation in a Patient With Schizophrenia. Front Psychiatry. 2020 Mar 17;11:174. doi: 10.3389/fpsyt.2020.00174. eCollection 2020. PMID 32256404
- [Background] Polinder S, Cnossen MC, Real RGL, Covic A, Gorbunova A, Voormolen DC, Master CL, Haagsma JA, Diaz-Arrastia R, von Steinbuechel N. A Multidimensional Approach to Post-concussion Symptoms in Mild Traumatic Brain Injury. Front Neurol. 2018 Dec 19;9:1113. doi: 10.3389/fneur.2018.01113. eCollection 2018. PMID 30619066
- [Background] Maas AIR, Menon DK, Adelson PD, Andelic N, Bell MJ, Belli A, Bragge P, Brazinova A, Buki A, Chesnut RM, Citerio G, Coburn M, Cooper DJ, Crowder AT, Czeiter E, Czosnyka M, Diaz-Arrastia R, Dreier JP, Duhaime AC, Ercole A, van Essen TA, Feigin VL, Gao G, Giacino J, Gonzalez-Lara LE, Gruen RL, Gupta D, Hartings JA, Hill S, Jiang JY, Ketharanathan N, Kompanje EJO, Lanyon L, Laureys S, Lecky F, Levin H, Lingsma HF, Maegele M, Majdan M, Manley G, Marsteller J, Mascia L, McFadyen C, Mondello S, Newcombe V, Palotie A, Parizel PM, Peul W, Piercy J, Polinder S, Puybasset L, Rasmussen TE, Rossaint R, Smielewski P, Soderberg J, Stanworth SJ, Stein MB, von Steinbuchel N, Stewart W, Steyerberg EW, Stocchetti N, Synnot A, Te Ao B, Tenovuo O, Theadom A, Tibboel D, Videtta W, Wang KKW, Williams WH, Wilson L, Yaffe K; InTBIR Participants and Investigators. Traumatic brain injury: integrated approaches to improve prevention, clinical care, and research. Lancet Neurol. 2017 Dec;16(12):987-1048. doi: 10.1016/S1474-4422(17)30371-X. Epub 2017 Nov 6. No abstract available. PMID 29122524
- [Background] Romero Lauro LJ, Rosanova M, Mattavelli G, Convento S, Pisoni A, Opitz A, Bolognini N, Vallar G. TDCS increases cortical excitability: direct evidence from TMS-EEG. Cortex. 2014 Sep;58:99-111. doi: 10.1016/j.cortex.2014.05.003. Epub 2014 Jun 6. PMID 24998337
- [Background] Jo JM, Kim YH, Ko MH, Ohn SH, Joen B, Lee KH. Enhancing the working memory of stroke patients using tDCS. Am J Phys Med Rehabil. 2009 May;88(5):404-9. doi: 10.1097/PHM.0b013e3181a0e4cb. PMID 19620953
- [Background] Dhaliwal SK, Meek BP, Modirrousta MM. Non-Invasive Brain Stimulation for the Treatment of Symptoms Following Traumatic Brain Injury. Front Psychiatry. 2015 Aug 26;6:119. doi: 10.3389/fpsyt.2015.00119. eCollection 2015. PMID 26379560
- [Background] Rushby JA, De Blasio FM, Logan JA, Wearne T, Kornfeld E, Wilson EJ, Loo C, Martin D, McDonald S. tDCS effects on task-related activation and working memory performance in traumatic brain injury: A within group randomized controlled trial. Neuropsychol Rehabil. 2021 Jun;31(5):814-836. doi: 10.1080/09602011.2020.1733620. Epub 2020 Mar 2. PMID 32114899
- [Background] Liebrand M, Karabanov A, Antonenko D, Floel A, Siebner HR, Classen J, Kramer UM, Tzvi E. Beneficial effects of cerebellar tDCS on motor learning are associated with altered putamen-cerebellar connectivity: A simultaneous tDCS-fMRI study. Neuroimage. 2020 Dec;223:117363. doi: 10.1016/j.neuroimage.2020.117363. Epub 2020 Sep 9. PMID 32919057
- [Background] Workman CD, Fietsam AC, Rudroff T. Different Effects of 2 mA and 4 mA Transcranial Direct Current Stimulation on Muscle Activity and Torque in a Maximal Isokinetic Fatigue Task. Front Hum Neurosci. 2020 Jun 25;14:240. doi: 10.3389/fnhum.2020.00240. eCollection 2020. PMID 32714170
- [Background] Antal A, Nitsche MA, Paulus W. Transcranial direct current stimulation and the visual cortex. Brain Res Bull. 2006 Feb 15;68(6):459-63. doi: 10.1016/j.brainresbull.2005.10.006. Epub 2005 Nov 2. PMID 16459203
- [Background] Hummel FC, Celnik P, Pascual-Leone A, Fregni F, Byblow WD, Buetefisch CM, Rothwell J, Cohen LG, Gerloff C. Controversy: Noninvasive and invasive cortical stimulation show efficacy in treating stroke patients. Brain Stimul. 2008 Oct;1(4):370-82. doi: 10.1016/j.brs.2008.09.003. Epub 2008 Oct 9. PMID 20633395
- [Background] Stagg CJ, Nitsche MA. Physiological basis of transcranial direct current stimulation. Neuroscientist. 2011 Feb;17(1):37-53. doi: 10.1177/1073858410386614. PMID 21343407
- [Background] Liebetanz D, Koch R, Mayenfels S, Konig F, Paulus W, Nitsche MA. Safety limits of cathodal transcranial direct current stimulation in rats. Clin Neurophysiol. 2009 Jun;120(6):1161-7. doi: 10.1016/j.clinph.2009.01.022. Epub 2009 Apr 28. PMID 19403329
- [Background] Workman CD, Fietsam AC, Rudroff T. Tolerability and Blinding of Transcranial Direct Current Stimulation in People with Parkinson's Disease: A Critical Review. Brain Sci. 2020 Jul 20;10(7):467. doi: 10.3390/brainsci10070467. PMID 32698528